CLINICAL TRIAL: NCT00001055
Title: A Phase I Safety and Immunogenicity Trial of Live Recombinant Canarypox ALVAC-HIV (vCP205) in HIV-1 Uninfected Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 022; 10572 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; Avipoxvirus; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: ALVAC-HIV MN120TMG (vCP205)
Biological: ALVAC-RG Rabies Glycoprotein (vCP65)
Biological: rgp120/HIV-1 SF-2

SUMMARY:
To evaluate the safety and immunogenicity of ALVAC-HIV MN120TMG (vCP205) in comparison to ALVAC-RG rabies glycoprotein (vCP65) as a control when administered in HIV-1 negative volunteers.

ALVAC-HIV vCP205 is a second generation candidate vaccine that can be used to induce a humoral and cellular response against several antigens. This recombinant construct is based on the canarypox vector termed ALVAC and expresses gp120 of the HIV MN strain, plus the transmembrane portion of the LAI strain as well as gag and protease.

DETAILED DESCRIPTION:
ALVAC-HIV vCP205 is a second generation candidate vaccine that can be used to induce a humoral and cellular response against several antigens. This recombinant construct is based on the canarypox vector termed ALVAC and expresses gp120 of the HIV MN strain, plus the transmembrane portion of the LAI strain as well as gag and protease.

Volunteers are randomized to receive doses of ALVAC-HIV vCP205 or ALVAC-HIV vCP65 control or both according to varying schedules over 12 months (was 6 months, amended 11/17/95) with a 12 month follow up. [AS PER AMENDMENT 5/29/98: One additional follow-up visit is required at 30-36 months.]

ELIGIBILITY:
Inclusion Criteria

Volunteers must have:

* Normal history and physical exam.
* Negative ELISA and Western blot for HIV.
* CD4 count >= 400 cells/mm3.
* Normal urine dipstick with esterase and nitrite.
* Occupational responsibilities that preclude compliance.

Exclusion Criteria

Co-existing Condition:

Volunteers with the following symptoms or conditions are excluded:

* Positive hepatitis B surface antigen.
* Medical or psychiatric condition (such as recent suicidal ideation or present psychosis) that precludes compliance.
* Active syphilis. NOTE: Subjects with serology documented to be a false positive or due to a remote (> 6 months) treated infection are eligible.
* Active tuberculosis. NOTE: Subjects with a positive PPD and a normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy are eligible.
* Allergy to egg products or neomycin.

Volunteers with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, autoimmune disease or use of immunosuppressive medications.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* Prior immunization against rabies.
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension).
* Prior psychiatric condition (such as history of suicide attempts or past psychosis) that precludes compliance.
* History of cancer unless there has been surgical excision that is considered to have achieved cure.
* Occupational responsibilities that preclude compliance.

Prior Medication:

Excluded:

* Live attenuated vaccines within 60 days prior to study entry. NOTE: Medically indicated killed or subunit vaccines (e.g., influenza, pneumococcal) do not exclude if administered at least 2 weeks from HIV immunizations.
* Experimental agents within 30 days prior to study entry.
* Prior HIV vaccines.
* Prior rabies immunization.

Prior Treatment:

Excluded:

* Blood products or immunoglobulin within 6 months prior to study entry.

Risk Behavior:

Excluded: Identifiable high-risk behavior for HIV infection, such as:

* injection drug use within past 12 months; higher- or intermediate-risk sexual behavior.
* Occupational exposure to birds. Low risk sexual behavior.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76
Dates: Study Completion 1997-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey L, Study Chair
Locations (6):
- United States (6):
  - UAB AVEG, Birmingham, Alabama
  - JHU AVEG, Baltimore, Maryland
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Ferrari G, Humphrey W, Corr K, Tartaglia J, Clements-Mann ML, Corey LC, Duliege AM, Excler JL, Weinhold KJ. Frequency and duration of HIV-1 specific cytolytic reactivities elicited in response to candidate AIDS vaccines. HIV Pathog Treat Conf. 1998 Mar 13-19:87 (abstract no 4026)
- [Background] Ferrari G, Humphrey W, McElrath MJ, Excler JL, Duliege AM, Clements ML, Corey LC, Bolognesi DP, Weinhold KJ. Clade B-based HIV-1 vaccines elicit cross-clade cytotoxic T lymphocyte reactivities in uninfected volunteers. Proc Natl Acad Sci U S A. 1997 Feb 18;94(4):1396-401. doi: 10.1073/pnas.94.4.1396. PMID 9037064
- [Background] Corey L, Weinhold K, Montefiori D, McElrath J, Excler JL, Duliege AM, Stablein D. Combination candidate HIV vaccines using a canarypox vector (vCP205) followed by boosting with gp120(SF-2). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:209 (abstract no LB18)
- [Background] Corey L, Weinhold K, McElrath J, Excler J-L, Duliege AM, Clements ML, Belshe R, Dolin R, Graham B. AVEU 022: safety and immunogenicity of live recombinant canarypox vector containing the envelope, gag and protease genes of HIV-1 in seronegative adult volunteers. Oral Abstract, 11th International Conference on AIDS, Vancouver, Canada, July 7-12, 1996 [Mo.A282]
- [Background] Kaslow RA, Rivers C, Goepfert P, Tang J, El Habib R, Weinhold K, Mulligan MJ. Association of HLA class I alleles with cytotoxic T-lymphocyte (CTL) responses to gag and env in recipients of ALVAC-HIV canarypox vaccines. 7th Conference on Retroviruses and Opportunistic Infections. 2000 Jan 30-Feb 2 [Poster 818]
- [Background] Egan MA, Pavlat WA, Tartaglia J, Paoletti E, Weinhold KJ, Clements ML, Siliciano RF. Induction of human immunodeficiency virus type 1 (HIV-1)-specific cytolytic T lymphocyte responses in seronegative adults by a nonreplicating, host-range-restricted canarypox vector (ALVAC) carrying the HIV-1MN env gene. J Infect Dis. 1995 Jun;171(6):1623-7. doi: 10.1093/infdis/171.6.1623. PMID 7769304
- [Background] Castillo RC, Arango-Jaramllo S, Humphrey W, Weinhold K, Schwartz DH. Vaccine induced CTL activity correlates with resistant phenotype in an in vitro challenge system. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:95 (abstract no 91)
- [Background] Sabbaj S, Corey L, Evans T, Keefer M, Excler JL, Duliege AM, Mulligan MJ, McGhee JR. Cytokine profiles in human PBMC T cell cultures stimulated with HIV antigens in seronegative volunteers immunized with canarypox expressing HIV antigens and boosted with recombinant SF2 GP120. Conf Adv AIDS Vaccine Dev. 1997 May 4-7:215 (Poster 110)
- [Background] Evans T, Corey L, Clements-Mann ML, Weinhold K, Belshe RB, Excler JL, Duliege AM. CD8+ CTL induced in AIDS vaccine evaluation group phase I trials using canarypox vectors (ALVAC) encoding multiple HIV gene products (vCP125, vCP205, vCP300) given with or without subunit boost. Int Conf AIDS. 1998;12:277 (abstract no 495/21192)
- [Background] Carruth LM, Greten TF, Murray CE, Castro MG, Crone SN, Pavlat W, Schneck JP, Siliciano RF. An algorithm for evaluating human cytotoxic T lymphocyte responses to candidate AIDS vaccines. AIDS Res Hum Retroviruses. 1999 Jul 20;15(11):1021-34. doi: 10.1089/088922299310539. PMID 10445814